CLINICAL TRIAL: NCT03521882
Title: Timed Interval Measurement of Eotaxin in Stroke Study
Acronym: TIMES
Status: Completed | Type: Observational
Sponsor: Royal Devon and Exeter NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: Protocol v5 15/05/17
Record Dates: First submitted 2018-04-30; First posted 2018-05-11 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Stroke, Acute
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stroke Symptom Participants
- Healthy Controls

SUMMARY:
Stroke is caused by sudden changes in blood flow in the brain. This can be fatal or can result in permanent disability. A fast diagnosis is essential to initiate effective interventions and optimize benefits to patients. There are other diseases that can look like a stroke and these are called "stroke mimics". The quicker that stroke mimics can be ruled out the faster a stroke can be diagnosed and treatment can be given. The investigators may be able to use chemicals in the blood to rapidly confirm that a person has had a stroke. One such chemical is called eotaxin. Eotaxin has been found to be changed in sufferers of a stroke but not in those with stroke mimics. However, more research is needed to confirm the usefulness of eotaxin. This feasibility study aims to provide the foundations to allow a large scale trial of this test. The study aims to recruit participants that have had a stroke or a stroke mimic from the Acute Stroke Unit and Stroke clinic at the Royal Devon and Exeter Hospital. Up to 6 blood samples will be taken from each participant at different times over one week. Eotaxin will be measured in these samples and in participant's leftover samples taken for clinical care. This is needed because the investigators know that the amount of eotaxin changes in the blood after a stroke but we do not know how quickly this change happens and for how long the change occurs. The study will also allow the investigators to understand how many participants will be needed for a large scale trial and the challenges that may be faced in recruiting participants.

ELIGIBILITY:
Inclusion Criteria:

* Presenting with focal neurological symptoms suggestive of stroke
* Aged over 18 years

Exclusion Criteria:

* Presenting later than 12 hours after symptom onset
* Under 18 years of age
* History of cardiovascular disease (Healthy Controls)
* History of neurological disease (Healthy Controls)
* History of stroke mimics (Healthy Controls)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals presenting to hospital with focal neurological symptoms suggestive of stroke aged over 18 years.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Primary Outcome | 0 to 7 days
  Plasma Eotaxin Concentration

CONTACTS AND LOCATIONS:
Overall Officials: Salim Elyas, PhD MRCP, Principal Investigator — Royal Devon and Exeter NHS Foundation Trust
Locations (1):
- Royal Devon & Exeter NHS Foundation Trust, Exeter, Devon, United Kingdom